CLINICAL TRIAL: NCT02467517
Title: Ketamine and Neuropathic Pain
Acronym: KETAPAIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0235
Record Dates: First submitted 2015-05-29; First posted 2015-06-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Ketamine; Magnesium sulfate; Quality of life; Anxiety and depression; Mood and sleep
MeSH Terms: conditions — Neuralgia; Anxiety Disorders; Depression | interventions — Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- INTRAVENOUS KETAMINE (Experimental)
  Interventions: Drug: Ketamine; Drug: Magnesium Sulfate; Drug: placebo : sodium chloride

INTERVENTIONS:
Drug: Ketamine
Drug: Magnesium Sulfate
Drug: placebo : sodium chloride

SUMMARY:
The primary outcome is to compare the analgesic efficacy of intravenous ketamine treatment to that of a placebo in patients with refractory neuropathic pain.

The secondary outcomes are:

1. - To compare the additive analgesic efficacy of prior administration of magnesium sulfate to that of placebo and ketamine only, on the effectiveness of intravenous ketamine treatment,
2. - To study the evolution time of pain and analgesia after the intravenous administration of ketamine and placebo,
3. - To study the correlation of the analgesic response to administered products respectively ketamine, ketamine and magnesium sulfate, placebo.

DETAILED DESCRIPTION:
Description of the study:

Single-center clinical trial, controlled, randomized, double-blind, crossover design, against inactive placebo.

Each patient will receive successively the 3 products (ketamine / placebo, ketamine / magnesium sulfate, placebo / placebo) follows a predeter randomization list, with a wash-out period between each administration.

Visit 1

-Inclusion visit, signature of informed consent form, clinical examination and fill questionnaires.

For women of childbearing age a pregnancy test will be performed.The pain will be measured by a numerical scale.

The pain will be evaluated by scoring on a numerical scale. A booklet for monitoring analgesic concomitant medication and overall pain on a numerical scale will be given to the patient 14 days before the programmed infusion.

Visit 2 : Period 1 Day 0

Clinical examination, return of booklet completed by patient and fill questionnaires.

The pain will be evaluated by scoring on a numerical scale before and after the infusion.

For women of childbearing age a pregnancy test will be performed. Treatment allocation period follows a predeter randomization list. At the end of the infusion, a booklet for monitoring will be given to patients for the following weeks in order to score their overall pain until the next study period.

The output of the hospital patient (CPC / CETD) after each treatment will be authorized by the investigator.

Wash-out period: 5 weeks.

Phone call 1 (Day 1):

Patients will be called by phone to collect adverse events and concomitant medications. If necessary, the patients should return to consult the CPC / CETD for a clinical examination.

Patients will be called the week before their scheduled visit, if at that time their spontaneous pain is still low, according to the opinion of the investigator, the infusion visit will be shifted to allow the pain level back its basal level.

Visit 3 : Period 2 : Day 36 +/- 3 days

Same of period 1.

Phone call 2 J 37 +/- 3 days:

Same of phone call 1.

Visit 4 : Period 3 : Day 72 +/- 3 days

Same of period 1

Phone call 3 J 73 +/- 3 days:

Same of phone call 1.

Visit 5 : Day 108 +/- 3 days

Clinical examination, return of booklet completed by patient and fill questionnaires.

The pain will be evaluated by scoring on a numerical scale For women of childbearing age a pregnancy test will be performed. This visit is the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient (s) are at least18 years old, with chronic pain (for more than 3 months), having the characteristics of a peripheral or central neuropathy, follow (s) at the Pain Clinic CHU Clermont-Ferrand and justifying the establishment of a therapeutic program including intravenous infusion of ketamine (as therapeutic test);
* Patient (s) who had never received ketamine infusion under the care of their neuropathic pain;
* History of illness compatible with an injury or disease of the somatosensory system;
* Localized pain in an anatomical neuro territory;
* Neurological examination shows sensory abnormalities,
* The patients of childbearing potential must use effective contraception throughout the study;
* For womens of childbearing age, they will be enrolled in the study after a negative urine pregnancy test; in case of suspicion of pregnancy, a blood pregnancy test should be performed;
* Cooperation and willing to follow the study;
* Acceptance to give written consent;
* Affiliated to the French social security;
* Inscription or acceptation of inscription in the national register of volunteers involved in trials.

Exclusion Criteria:

* Patient (s) who have received intravenous ketamine infusion;
* Patients with one or many contraindication to ketamine administration: known hypersensitivity to ketamine in which one of the constituents of the product, uncontrolled high blood pressure, severe cardiac insufficiency;
* Patients with one or many contraindication of magnesium sulfate administration: Patients with severe renal impairment;
* Patients with one or many contraindication to administration of sodium chloride: water inflation, fluid retention;
* Patients with a medical history and / or surgical judged by the investigator to be not consistent with the clinical trial;
* Patients with drug treatments judged by the investigator to be not consistent with the clinical trial;
* Pregnancy or lactation women;
* Patient who participated in another clinical trial, located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial;
* Patients with cooperation and understanding not to adhere strictly to the conditions provided in the clinical trial;
* Patients receiving a measure of legal protection (guardianship…);
* Patients are not affiliated to the System of the French Social Security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | at day 1 and for a period of 5 weeks (35 days).

SECONDARY OUTCOMES:
Intensity of the average | at day 1
  Intensity of the average daily pain evaluated by a numerical rating scale (NRS) assessed using a booklet
Intensity of maximum daily pain | at day 1
  Intensity of maximum daily pain evaluated by a numerical rating scale (NRS) assessed using a booklet,
Impact on quality of life | at day 1
  Impact on quality of life, mood and sleep assessed by questionnaires.
Impact on mood | at day 1
  Impact on quality of life, mood and sleep assessed by questionnaires.
Impact on sleep | at day 1
  Impact on quality of life, mood and sleep assessed by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France